CLINICAL TRIAL: NCT04110756
Title: Promoting Adolescent Health Behavior Change With Clinically Integrated Sample-Efficient Policy Gradient Methods
Brief Title: ChangeGradients: Promoting Adolescent Health Behavior Change
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: North Carolina State University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-28893; R01CA247705 (NIH)
Record Dates: First submitted 2019-09-10; First posted 2019-10-01 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Drinking; Self Efficacy; Adolescent Behavior; Risk-Taking; Cancer
Keywords: Alcohol- Prevention/Control; Adolescent behavior; Video games- psychology
MeSH Terms: conditions — Alcohol Drinking; Adolescent Behavior; Risk-Taking; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (ChangeGradients) (Experimental): Adolescent participants will be introduced to the intervention through a brief introductory video trailer during their clinic visit and receive a link that enables them to engage with CHANGEGRADIENTS interactive narratives at home over a course of four weeks (i.e., one per week) on a personal computing device (e.g., laptop or tablet).
  Interventions: Behavioral: ChangeGradients
- No Intervention (Usual Care) (No Intervention): Participants will receive usual care at the clinic.

INTERVENTIONS:
Behavioral: ChangeGradients — CHANGEGRADIENTS is an interactive web-based tool which includes narrative-centered behavior change experiences that are dynamically generated.
  Other Names: CHANGEGRADIENTS system
  Arms: Treatment (ChangeGradients)

SUMMARY:
As most adolescents visit a healthcare provider once a year, health behavior change interventions linked to clinic-based health information technologies hold significant promise for improving healthcare quality and subsequent behavioral health outcomes for adolescents (Baird, 2014, Harris, 2017). Recognizing the potential to leverage recent advances in machine learning and interactive narrative environments, the investigators are now well positioned to design health behavior change systems that extend the reach of clinicians to realize significant impacts on behavior change for adolescent preventive health.

The proposed project centers on the design, development, and evaluation of a clinically-integrated health behavior change system for adolescents. CHANGEGRADIENTS will introduce an innovative reinforcement learning-based feedback loop in which adolescent patients interact with personalized behavior change interactive narratives that are dynamically personalized and realized in a rich narrative-centered virtual environment. CHANGEGRADIENTS will iteratively improve its behavior change models using policy gradient methods for Reinforcement Learning (RL) designed to optimize adolescents' achieved behavior change outcomes. This in turn will enable CHANGEGRADIENTS to generate more effective behavior change narratives, which will then lead to further improved behavior change outcomes. With a focus on risky behaviors and an emphasis on alcohol use, adolescents will interact with CHANGEGRADIENTS to develop an experiential understanding of the dynamics and consequences of their alcohol use decisions. The proposed project holds significant transformative potential for (1) producing theoretical and practical advances in how to realize significant impacts on adolescent health behavior change through novel interactive narrative technologies integrated with policy-based reinforcement learning, (2) devising sample-efficient policy gradient methods for RL that produce personalized behavior change experiences by integrating theoretically based models of health behavior change with data-driven models of interactive narrative generation, and (3) promoting new models for integrating personalized health behavior change technologies into clinical care that extend the effective reach of clinicians.

DETAILED DESCRIPTION:
STUDY AIMS:

I. Design, develop, and iteratively refine a policy-based reinforcement learning behavior change system for preventive adolescent health (Part 1).

II. Investigate the impact of a clinically integrated sample-efficient policy gradient-based behavior change system on adolescent behavior (Part 2).

The project will culminate with an investigation of the behavioral effects of the CHANGEGRADIENTS system using adolescent patients recruited from two outpatient primary care clinics within the UCSF Department of Pediatrics: Mt. Zion Pediatrics and the Adolescent/Young Adult Clinic. It is hypothesized that adolescents who interact with CHANGEGRADIENTS will reduce number of days of alcohol use, reduce binge drinking, and increase self-efficacy to engage in healthy behavior and avoid risky substance use.

It is anticipated that CHANGEGRADIENTS will provide a testbed for a broad range of health behavior change research and serve as the foundation for next generation personalized preventive healthcare through computationally enabled behavior change that is designed to be tightly integrated into clinical practice workflow. By taking advantage of the high degree of adaptive interactivity offered by its personalized behavior change environment, CHANGEGRADIENTS holds significant potential for creating compelling interactions that promote self-efficacy and engagement in healthy lifestyle behaviors to prevent cancer through improving cancer-related behaviors and risk factors.

PART 1 of the study (Focus Group) has closed to enrollment.

PART 2 of the study (Randomized Clinical Trial) is planned for enrollment upon finalization of data collected in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 15 and 17 years of age
* Report current alcohol use
* Presenting for a well-visit at UCSF Pediatric primary care clinics (the Mt. Zion Pediatric Primary Care Practices at UCSF and The Adolescent/Young Adult Clinic at UCSF)

Exclusion Criteria:

* Non-English speakers

Ages: 15 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-02-12 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Mean scores on assessment of Alcohol Use | 30 days
  Standard validated questions taken from the "Alcohol and other Drug Use" scale of the Youth Risk Behavior Surveillance Survey (CDC surveillance system that monitors adolescent risk behavior) will be administered. Measures include quantity and frequency of use and safety (drinking and driving), Current use of alcohol measured by quantity and frequency of use in the past 30 days (Centers for Disease Control and Prevention, 2018). Scale ranges vary based on questions and questions are scored individually. Responses to questions about alcohol use in general (past 12 months and ever) are scored as No = 0 and Yes = 1. Values on questions about alcohol use in the past 30 days are scored on a scale from 0-7, with higher values corresponding to greater alcohol consumption. Questions about drinking and driving are scored on a scale from 0-5 with higher numbers corresponding to more frequent instances of driving/being driven by others after alcohol was consumed.
Mean score on a Self-efficacy tool developed by Drs Elizabeth Ozer and Dr. Albert Bandura | 30 days
  Self-efficacy will be measured using a tool developed by Drs Elizabeth Ozer and Dr. Albert Bandura designed for this study. The tool assesses confidence in avoiding drinking in various scenarios. Participants are asked to rate level of confidence in drinking avoidance across various situations. Responses are rated on a scale of 0 to 10, with a rating of 0 indicating 'not at all confident', a rating of 5 indicating 'moderately confident', and rating of 10 indicating t 'completely confident'. Scenarios include: "When a close friend offers you a drink," and, "When you feel depressed or nervous." Scores on this assessment are calculated by summing participant responses and dividing by the number of questions to obtain a mean self-efficacy score.
Quality of Care: Adolescent Report of the Visit (AROV) | 1 day, immediately following baseline clinic visit
  The Adolescent Report of the Visit (AROV) is a validated measure to assess the quality of care delivered to adolescents (Ozer, 2004), which has been utilized in clinics nationally and internationally (Sanci, 2015). The investigators are specifically using questions from this measure assessing provider rates of screening and counseling adolescents for alcohol use during adolescent visits. All questions are scored separately on a binary scale, with response scoring as No = 0 and Yes = 1. An answer of Yes to any item indicates higher quality of care.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ozer, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco Adolescent and Young Adult Medicine Clinic, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared with research collaborators during the course of the study
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Baird A, Nowak S. Why primary care practices should become digital health information hubs for their patients. BMC Fam Pract. 2014 Nov 25;15:190. doi: 10.1186/s12875-014-0190-9. PMID 25421733
- [Background] Harris SK, Aalsma MC, Weitzman ER, Garcia-Huidobro D, Wong C, Hadland SE, Santelli J, Park MJ, Ozer EM. Research on Clinical Preventive Services for Adolescents and Young Adults: Where Are We and Where Do We Need to Go? J Adolesc Health. 2017 Mar;60(3):249-260. doi: 10.1016/j.jadohealth.2016.10.005. Epub 2016 Dec 20. PMID 28011064
- [Background] Ozer EM, Bandura A. Mechanisms governing empowerment effects: a self-efficacy analysis. J Pers Soc Psychol. 1990 Mar;58(3):472-86. doi: 10.1037//0022-3514.58.3.472. PMID 2324938
- [Background] Ozer EM, Adams SH, Orrell-Valente JK, Wibbelsman CJ, Lustig JL, Millstein SG, Garber AK, Irwin CE Jr. Does delivering preventive services in primary care reduce adolescent risky behavior? J Adolesc Health. 2011 Nov;49(5):476-82. doi: 10.1016/j.jadohealth.2011.02.011. Epub 2011 Jun 8. PMID 22018561
- [Background] Sanci L, Chondros P, Sawyer S, Pirkis J, Ozer E, Hegarty K, Yang F, Grabsch B, Shiell A, Cahill H, Ambresin AE, Patterson E, Patton G. Responding to Young People's Health Risks in Primary Care: A Cluster Randomised Trial of Training Clinicians in Screening and Motivational Interviewing. PLoS One. 2015 Sep 30;10(9):e0137581. doi: 10.1371/journal.pone.0137581. eCollection 2015. PMID 26422235
- [Background] Ozer EM, Adams SH, Lustig JL, Millstein SG, Wibbelsman CJ, Babb J. The effect of preventive services on adolescent behavior (abstract). Pediatric Research. 2004;53(suppl. 4, pt. 2):265A.
- [Background] Ozer EM. The impact of childcare responsibility and self-efficacy on the psychological health of working mothers. Psychology of Women Quarterly. 1995;19:315-35.
- [Background] Ozer E, Rowe J, Tebb K, Culbertson K, Berna M, Jasik C, et al. A self-adaptive personalized behavior change system for adolescent preventive care. The Indian Journal of Pediatrics, Special Supplement The International Association for Adolescent Health, 11th World Congress on Adolescent Health, 27-29 October, 2017, New Delhi, India2017. p. SS-1.
- See also: Facts About Underage Drinking- National Institute on Alcohol Abuse and Alcoholism — https://www.niaaa.nih.gov/publications/brochures-and-fact-sheets/underage-drinking

DOCUMENTS (1):
  • Informed Consent Form (2023-08-24): https://cdn.clinicaltrials.gov/large-docs/56/NCT04110756/ICF_000.pdf